CLINICAL TRIAL: NCT05150509
Title: Association of Salivary Amino Acid With Oral Squamous Cell Carcinoma Identified by Liquid Chromatography Mass Spectroscopy
Brief Title: Association of Salivary Amino Acid Level With OSCC Identified By Liquid Chromatography Mass Spectroscopy
Acronym: OSCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DR. MALA KHAN (Other Government)
Collaborators: Bangladesh Reference Institute of Chemical Measurements (BRICM) (Other Government)
Responsible Party: Sponsor-Investigator, DR. MALA KHAN, Chief Scientific Officer, Bangladesh Reference Institute of Chemical Measurements (BRICM)
Organization: Bangladesh Reference Institute of Chemical Measurements (BRICM) (Other Government)
Other Study IDs: ORAL SQUAMOUS CELL CARCINOMA
Record Dates: First submitted 2021-10-25; First posted 2021-12-09 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Oral saliva is collected for the intervention purpose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Progressive Disease and without Progressive Disease: 1. Patients with Progressive Disease Patients with metastasis and/or recurrent OSCC were considered as a group of subjects with progressive disease.
  2. Patients with without Progressive Disease Patients without metastasis and/or recurrent OSCC were considered as a group of subjects without progressive disease.
  Interventions: Diagnostic Test: Oral Squamous Cell Carcinoma

INTERVENTIONS:
Diagnostic Test: Oral Squamous Cell Carcinoma — To identify the association of elevated level of specific amino acids in OSCC by Liquid Chromatography Mass Spectrometry

SUMMARY:
Oral Squamous Cell Carcinoma (OSCC) is the most common oral malignancy worldwide. The prognosis of the OSCC patient is not significant despite the modern treatment facilities. Late presentation is one of the most crucial cause of this and for that reason, the importance of early diagnosis of OSCC should be the main concern. Till now, incisional biopsy followed by histopathological examination is the gold standard for diagnosis of oral cancer. The aim of the present study is to find out the association of salivary amino acid levels with oral squamous cell carcinoma, whether the levels are increased or decreased in the patient suffering from OSCC. This might be helpful for early diagnosis of oral cancer and better prognosis.

DETAILED DESCRIPTION:
1. Introduction:

   Oral cancer is an abnormal growth of tissue, originates from the tissue in and around the mouth which is uncoordinated with that of the surrounding normal tissue. Among all oral cancers, oral squamous cell carcinoma (OSCC) is the most common (90%) malignant epithelial neoplasm of the oral cavity. It is an alarming public health problem in the world due to its prevalence, high incidence rate and mortality. According to the recent data of GLOBOCAN 2020, 377713 newly diagnosed lip and oral cavity squamous cell carcinoma patients diagnosed worldwide which is about 2% of all cancer reported. Oral squamous cell carcinoma (OSCC) is the 6th most common cancer worldwide. Recent global reports suggest that the largest portion of the reported cases are from Asia (65.8%), but in the South Asia region, oral cancer is the 3rd most common cancer. One of the critical factor of the high mortality rate of OSCC is that initially many of the lesion is asymptomatic. As a result, they come at the late stage of the disease to the physician and ultimately have a poor prognosis. Research showed that, when an OSCC is in stage I, the 5-year survival rate is 80% but it drops to 20-40% when the disease is in stage IV. For the diagnosis of OSCC, after the initial clinical examination, incisional biopsy followed by histopathological examination is still considered as a gold standard, but the method has many limitations. Invasive procedure needs special expertise for taking biopsy sample from the representative areas and need expert histopathologist for confirmation. Moreover, taking a tissue sample from behind the visible area such as the base of the tongue, posterior pillar and incase of restricted jaw opening is very difficult or sometimes impossible.

   Human saliva is the secretion from three major salivary gland parotid, submandibular, sublingual and numerous minor glands lie just beneath the mucosa of the oral cavity. It consists of water (99.5%), inorganic salts and enzymes (0.2%) and proteins (0.3%). It is helpful for the diagnosis of periodontitis, diabetes mellitus, HIV, dengue, mumps even breast cancer, pancreatic cancer, gastric cancer, lung cancer and oral cancer. Additionally, taking saliva samples has many advantages. Taking saliva is easier, and needs no invasive procedure or expertise. Besides, it has a sufficient amount of production and can be taken by the patient himself making the sample taking procedure cheaper. Salivary amino acids are the important metabolites for the diagnosis of a cancer patient. Amino acid is the raw product of protein synthesis. For this, when a cancer patient passes through a hypermetabolic and hypercatabolic state, there is a chance of protein imbalance. As the investigators know that amino acids are the byproducts of protein, it can give us a hint for the state of imbalance due to any cancer including oral squamous cell carcinoma. In addition, changes in amino acid concentration in the body fluid of cancer patient is significant according to several studies Mass spectrometry is a currently used platform for proteomics or metabolomics in biomedical research. Like other spectrometry method such as gas chromatography-mass spectrometry (GC-MS), capillary electrophoresis-mass spectrometry(CE-MS), two-dimensional electrophoresis mass spectrometry (2DE-MS), matrix-assisted laser desorption ionization-time of flight mass spectrometry (MALDI-TOF) and surface enhanced laser desorption ionization time-of-flight mass spectrometry (SELDI-TOF), Liquid chromatography-mass spectrometry (LC-MS) is widely used nowadays. It allows a quick and efficient separation and characterization of analytes in a given sample. Thus, it can help in rapid diagnosis of any disease by automated analysis of amino acid profiles with minimum effort and expenses. Many studies were conducted using LC-MS machine for saliva analysis for the diagnosis of several diseases and found significant results. To the best of my knowledge, very few studies were done to find out the salivary amino acid level from the patient having suspected oral lesion by LC-MS. Moreover, no study was performed for oral lesion diagnosis by analysis of amino acid profile using LC-MS in Bangladesh. The aim of this study is to find out the association of specific salivary amino acid levels with the patient of OSCC by Liquid Chromatography-Mass Spectrometry (LC-MS).
2. Rationale:

   OSCC is the 6th most common cancer worldwide, but in Asia the largest portion was reported recently and in South-east Asia, it is the 3rd most common cancer. Poor socio-economic condition, lack of consciousness and widely use of tobacco, betel quid chewing and alcohol intake are the main factors behind this. Research showed that early diagnosis of cancer reduces the mortality rate and hence can improve the treatment outcome. As a result, scientists are trying to find out an easy, quick and reliable method of diagnosis of OSCC.

   Although scalpel (incisional) biopsy followed by histopathological examination is still the gold standard for the diagnosis of the oral lesion but in the case of behind the visible area and in restricted mouth opening it is very difficult to collect the representative specimen. Moreover, the procedure is invasive and needs special equipment and expertise. In this aspect, to avoid the risk of invasive procedures and pain, body fluid analysis is the area of interest of the researcher nowadays.

   Among the other body fluid, saliva is very easy to collect, non-invasive and might have the property to diagnose of OSCC because it remains with the contact with the lesion. It has plenty of flow and less costly than the others.

   LC-MS machine is now widely used for metabolomics analysis all over the world. It has the capacity to analyze a sample more effectively and within a very short time. Measuring the amino acid and other components from the saliva can easily be done by this method. Due to some diseases, amino acid concentration of body fluid differs according to several studies. The investigators believe that for the Bangladeshi population there are significant associations between several salivary amino acid levels and OSCC, which can be identified by LC-MS.
3. General objective:

   To find out the association of salivary amino acid levels with oral squamous cell carcinoma (OSCC) identified by liquid chromatography-mass spectrometry.
4. Place of study:

   Oral and Maxillofacial Surgery Department, Bangabandhu Sheikh Mujib Medical University (BSMMU)and Bangladesh Reference Institute for Chemical Measurements (BRICM), Science lab, Dhanmondi, Dhaka.
5. Study Population:

   Patients and their attendants attending in outdoor and indoor clinic of Oral and Maxillofacial Surgery Department, BSMMU according to inclusion and exclusion criteria. Total sample size will be 110 and 55 in each group. Cases are the oral squamous cell carcinoma patients confirmed by incisional biopsy and controls are the relatively same age group and healthy individuals.
6. Study sample:

   Patients attending to the Department of Oral & Maxillofacial Surgery, histo-pathologically diagnosed as oral squamous cell carcinoma who will fulfill the selection criteria will be selected as cases. Control subjects will be taken from healthy individuals among the attendants of patients almost from the same age group of cases maintaining the inclusion criteria. The participants are classified into two goups Group A (Cases): Study group consists of 55 patients those having histopathologically confirmed Oral Squamous Cell Carcinoma (OSCC) Group B (Controls): This group consists of 55 healthy individuals with nothaving any history of cancer and without severe periodontal problems and dental caries.
7. Study variables:

   * Histopathology report
   * Level of salivary Amino acids detected by Liquid chromatography-mass spectrometry (LC-MS)
8. Ethical consideration:

   Ethical clearance for the study will be taken from the Institutional Review Board (IRB) of BSMMU prior to the commencement of this study. After the research protocol is approved by the committee, permission for the study will be taken from the Department of Oral and Maxillofacial Surgery, Bangabandhu Sheikh Mujib Medical University.

   The aims and objectives of the study along with its procedure, risks, stages and benefits of this study will be explained to the study subjects in an easily understandable local language. They will be assured that the risk of this research is minimum. But, this risk will be properly addressed by specialist doctor. If any problem arises related to the biopsy procedure or due to any step of this research activity, they will get the whole treatment in free of cost. During and after research program confidentiality would be maintained strictly. An ID number will be given to them and that will be helpful to the research program. All the papers belong to this ID number will be locked in office. Personal matter will not be used for analysis, producing article and release. Only the involved investigator will know all these and nobody will get their information.

   Their participation in this research program is absolutely voluntary. They can either deny participation or leave the research program at any time. That will not affect their treatment process. Their legal right will not be harmed by signing the consent form. A written informed consent will be taken from all the study subjects without exploiting any of their weakness. All the study subjects will be assured about their confidentiality and freedom to withdraw themselves from the study at any time.
9. Implementation of results:

   The result might be helpful to find out the association betweensalivary amino acidlevelsand oral squamous cell carcinoma (OSCC) patients. Thus, might be helpful in early detection of OSCC.

   The data will be helpful for future research and that will be considered baseline information for public health department.
10. Aim and Procedure:

The aim of the study is to find out the association of salivary amino acid levels with oral squamous cell carcinoma (OSCC).The study will be conducted at Oral and Maxillofacial Surgery Department of Bangabandhu Sheikh Mujib Medical University Patient with histologically confirmed OSCC will be enrolled as cases in the study by purposive convenient sampling technique to achieve the desired number. Approximately same number of the healthy individuals will be taken as control group for comparison. Then the saliva will be taken from the OSCC patient and from the control group. After taking in the sterile container and ensuring proper environment saliva sample will be carried to Designated Reference Institute for Chemical Measurements (DRICM), Science lab, Dhanmondi for analysis by liquid chromatography-mass spectrometry (LC-MS) machine. By this machine, the levels of 6 specific amino acids (Alanine, Valine, Glycine, Phenylalanine, Isoleucine, Lysine) will be measured. The data obtained from each individual will be recorded in predesigned data collection sheet separately. If participents are agreeing to participate in this research program, the responsible doctor will inform the participents in detail.

ELIGIBILITY:
Inclusion criteria for case

* Age: 18-70 years.
* Both genders.
* Patient with histo-pathologically diagnosedoral squamous carcinoma
* Willing to participate in the study. Inclusion criteria for controls
* Healthy patients without any malignancy
* Patients relatively almost the same age group of cases

Exclusion criteria for cases

* Patients with severe periodontitis and multiple carious teeth.
* Patients having other systemic diseases and cancer.
* Patients who cannot fulfill the inclusion criteria. Exclusion criteria for controls
* Having severe periodontal problemsor dental caries
* Suffering from any cancer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and their attendants attending in outdoor and indoor clinic of Oral and Maxillofacial Surgery Department, BSMMU according to inclusion and exclusion criteria. Total sample size will be 110 and 55 in each group. Cases are the oral squamous cell carcinoma patients confirmed by incisional biopsy and controls are the relatively same age group and healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study to establish a diagnostic test in the early detection of OSCC. | From December,2020 to February, 2022
  1. Total 110 samples, 55 in each group (case and control) will be included in the study and a questionnaire will be filled up by each participant based on their sociodemographic characteristics, personal habit and also the tumor staging of confirmed cancer cases.
  Saliva metabolite profiling of six amino acids (Alanine, Valine, Glycine, Phenylalanine, Isoleucine, Lysine) will be performed using LCMS/MS system.
  During metabolite profiling experiments, centroid data will be acquired for each sample from 50 to 1000 Da with a 0.10-sec scan time and a 0.01-sec interscan delay over an 18-min analysis time.
  3. The LCMS/MS data of OSCC and control saliva samples will be analyzed to identify potential discriminant variables. Selecting the method, investigator will create dataset, Researcher would like to (i) detect Peaks and (ii) collect markers. The investigators can create dataset display, and at this point, it is also possible to automatically print data into a text file.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dipayan Mojumder, BDS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (2):
- Bangladesh (2):
  - Bangladesh Reference Institute for Chemical Measurements, Dhaka, Dhanmondi
  - Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT05150509/ICF_000.pdf